CLINICAL TRIAL: NCT03816410
Title: Influence of Left Atrial Appendage Amputation on Natriuretic Peptides - a Randomized Controlled Trial
Brief Title: Natriuretic Peptides After Left Atrial Appendage Amputation
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Giessen (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Screening
Other Study IDs: SR-345-DP
Record Dates: First submitted 2019-01-22; First posted 2019-01-25 (Actual); Last update posted 2019-01-25 (Actual); Status verified 2019-01

CONDITIONS: Atrial Fibrillation
MeSH Terms: conditions — Atrial Fibrillation

STUDY DESIGN:
Intervention Model Description: 1:1 Randomization
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- LAA amputation group (Experimental)
  Interventions: Procedure: LAA amputation
- No LAA amputation group (No Intervention)

INTERVENTIONS:
Procedure: LAA amputation — complete surgical amputation of the left atrial appendage
  Arms: LAA amputation group

SUMMARY:
Surgical amputation of the left atrial appendage (LAA) is an established intervention during surgical atrial fibrillation (AF) therapy. However, its effects on the endocrine function of the left atrium are unclear. This study aims to quantify the serum levels of natriuretic peptides in patients who undergo concomitant surgical AF ablation with or without LAA amputation.

ELIGIBILITY:
Inclusion Criteria:

* Indication for concomitant AF therapy during cardiac surgery with cardiopulmonary bypass

Exclusion Criteria:

* Lack of informed consent

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 21 (Actual)
Dates: Start 2015-05-01 (Actual); Primary Completion 2015-10-30 (Actual); Study Completion 2018-12-01 (Actual)

PRIMARY OUTCOMES:
Serum levels of proANP and BNP until 800days post surgery | 800days

CONTACTS AND LOCATIONS:
Locations (1):
- Department of Adult and Pediatric Cardiovascular Surgery, Giessen, Germany

IPD SHARING:
Plan to Share IPD: No